CLINICAL TRIAL: NCT01344655
Title: A Single-centre, Double-blind, Double-dummy, Randomised, Crossover Study to Investigate the Effect of Formoterol HFA-pMDI Versus Salmeterol HFA-pMDI on Small Airways Physiological Parameters in COPD Patients
Brief Title: Study to Investigate the Effect of Formoterol vs Salmeterol on Small Airways Physiological Parameters in COPD Patients
Acronym: Imperial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0901-PR-0012; 2008-008656-16 (EudraCT Number)
Record Dates: First submitted 2010-11-29; First posted 2011-04-29 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formoterol 12 μg pMDI (Atimos®) (Experimental)
  Interventions: Drug: Atimos®
- Salmeterol 25 µg pMDI HFA (Serevent™) (Active Comparator)
  Interventions: Drug: Serevent™
- Matched Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atimos® — Formoterol 12 μg pMDI
  Arms: Formoterol 12 μg pMDI (Atimos®)
Drug: Serevent™ — Salmeterol 25 µg pMDI
  Arms: Salmeterol 25 µg pMDI HFA (Serevent™)
Drug: Placebo — placebo
  Arms: Matched Placebo

SUMMARY:
This is a crossover Study to investigate the effect of Formoterol versus Salmeterol on small airways physiological parameters in COPD patients.

DETAILED DESCRIPTION:
A Single-centre, Double-blind, Double-dummy, Randomised, Crossover Study to investigate the effect of Formoterol HFA-pMDI versus Salmeterol HFA-pMDI on small airways physiological parameters in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of COPD
* Post bronchodilator FEV1 between 30% and 80% predicted values at screening
* Post-bronchodilator FEV1/FVC < 0.7

Exclusion Criteria:

* Positive FEV1 reversibility test: FEV1 change greater than 200 mL and 12%
* History of another medical condition contraindicating participation in the study
* Clinical evidence of heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Respiratory Impedance by Impulse oscillometry | from 5 minutes to 8 hours post dose

SECONDARY OUTCOMES:
Exhaled Nitric Oxide | from 30 minutes to 8 hours post dose
Multiple Breath Nitrogen Washout | from 30 minutes to 8 hours post dose
Forced Expiratory Volume in the 1st second | from 30 minutes to 8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Omar S Usmani, MD, Principal Investigator — Imperial College London
Locations (1):
- Airway Disease Section, NHLI, Imperial College London, London, United Kingdom

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2008-008656-16